CLINICAL TRIAL: NCT02431546
Title: A Lifestyle-Based Mobile Health Strategy for Cardiovascular Disease Prevention in Graduates From Cardiac Rehabilitation: VIDA Pilot Study
Brief Title: VIDA Mobile Health Cardiovascular Prevention Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Vida Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00057493
Record Dates: First submitted 2015-04-28; First posted 2015-05-01 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Coronary Artery Disease
Keywords: Cardiology; Vascular; CAD; Duke; Cardiac Rehabilitation; Prevention; CVD; Mobile Health; Exercise
MeSH Terms: conditions — Coronary Artery Disease; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mobile Health Application Group (Experimental): VIDA is a mobile technology that is well positioned to provide healthcare coaching. After completing the CR program, each participant will have access to the VIDA mobile phone platform for the 12-week intervention, and be instructed to download the app on his/her smart phone. VIDA will assign an individual professional health coach selected from a pool of well-trained and experienced health professionals-nutritionists, fitness trainers, nurses and health educators. Each coach will engage their patient in a productive and meaningful health mentorship on a daily basis. The coach and patient work as a team to successfully set goals and make small changes that add up to significant improvements in the patients' dietary choices, physical activity, medication management, as well as understanding of their health status.
  Physical Activity: A goal of "total number of steps" to attain daily will be provided by the Duke study team to the patient and monitored using a Fitbit activity tracker.
  Interventions: Behavioral: Mobile Health Application
- Usual Care Group (No Intervention): Participants randomized to the usual care control arm will follow standard care as ordered by their individual, treating physician. Participants in the UC control arm will not receive any specific lifestyle recommendations from study personnel. They may, however, receive any lifestyle recommendations deemed appropriate by their usual clinical care providers. All participants will be contacted by study personnel in order to schedule visits at baseline and 12-weeks for the outcome assessments.

INTERVENTIONS:
Behavioral: Mobile Health Application — Health coaching is an innovative, holistic approach oriented towards one's full health and wellbeing. Coaches provide mentoring and support regarding many areas of life that impact one's health with a focus on skill-building. Health coaches do not provide medical advice, treat any medical conditions, provide mental health therapy, or provide individualized assessments of nutrient needs. Health coaches will not conduct medication counseling activities that would alter the prescribed regimen nor provide medication information/advice that would be considered the practice of medicine or pharmacy.
  A Fitbit activity monitor will be used to track daily physical activity and provide real-time feedback to the participant.
  Other Names: Health Coaches; Physical Activity Tracker
  Arms: Mobile Health Application Group

SUMMARY:
The purpose of this study is to understand the effects of a mobile health cardiovascular prevention program in patients who have recently graduated from cardiac rehabilitation. The mobile health program will focus on promoting healthy lifestyles through the use of a mobile application (app), mobile physical activity monitor and a system of remote health coaching.

By testing a novel mHealth intervention focused on lifestyle modification, this trial will address a critical evidence gap in the care of patients after they graduate from CR. Many patients who graduate from traditional CR struggle with unhealthy lifestyles, and these patients currently have no lifestyle-based care strategies to help them. The results of this study have the potential to lead to new sustainable and resource-efficient, lifestyle-based preventive care strategies for patients with stable CVD.

DETAILED DESCRIPTION:
This is a single-center, randomized trial designed to examine the hypothesis that a lifestyle-based mobile health cardiovascular disease (CVD) prevention program administered to graduates of a cardiac rehabilitation (CR) program will improve physical activity, body composition, fitness, and quality of life (QOL).

The investigators may enroll up to 52 men and women volunteers from a pool of graduates of the Duke Cardiac Rehabilitation Program who are initially eligible to participate in this study. Of the 52 men and women volunteers who may be initially consented, it is anticipated that a portion (potentially 30%) may drop out during the study timeline, and approximately 40 are expected to complete this study. Following informed consent and baseline testing, the participants will be randomized in a 3:1 fashion to receive VIDA's 12-week mHealth program focused on lifestyle modification through remote health coaching in order to improve physical activity, body composition, and fitness. The multi-domain mHealth intervention will mirror traditional CR programs by focusing primarily on a structured physical activity intervention within the context of a comprehensive lifestyle program. Physical activity will be monitored by Fitbits and will be integrated into VIDA's mHealth platform which will also include modules on physical activity, weight management, heart healthy diet, medication adherence, coping with a chronic disease, psychosocial management, and stress management/sleep. Health coaches will be used to guide patients through the 12-week program. All participants will undergo measures of physical activity, body composition, fitness, and QOL at baseline and at 12-weeks.

ELIGIBILITY:
Inclusion Criteria:

* Graduates of CR, who were originally enrolled in CR following myocardial infarction (MI), percutaneous coronary intervention (PCI), or coronary artery bypass graft (CABG) or with stable angina
* Adequate clinical stability has been achieved in the judgment of the investigator to allow participation in study assessments and the intervention
* Ability to participate in a mobile health program with access to smartphones utilizing Apple and Android platforms
* Signed informed consent document indicating that the patient understands the purpose of and procedures required for the study and is willing to participate in the study

Exclusion Criteria:

* Acute symptoms of coronary artery disease
* Decompensated heart failure
* Severe valvular heart disease
* Severe pulmonary hypertension
* End stage renal disease
* Heart failure, New York Heart Association (NYHA) class IV
* Cardiac transplantation
* Terminal illness with life expectancy < 1 year
* Impairment from stroke, injury or other medical disorder that precludes participation in the intervention
* Dementia that precludes ability to participate in and follow study protocols
* Enrollment in a clinical trial not approved for co-enrollment
* Inability or unwillingness to comply with the study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-07; Primary Completion 2017-03-20 (Actual); Study Completion 2017-03-20 (Actual)

PRIMARY OUTCOMES:
Change in fitness (peak VO2mL/kg/min) as measured by cardiopulmonary exercise test (CPET). | Baseline and 14-weeks
  peak VO2mL/kg/min

SECONDARY OUTCOMES:
Understand the feasibility and implementation of this novel mhealth treatment strategy. | 14-weeks
  Patient Satisfaction Survey
Change in Physical Activity as measured using a Fitbit | Baseline and 14-weeks
  Total number of steps, distance traveled and floors climbed.
Change in Quality of Life (QOL) as measured by Seattle Angina Questionnaire (SAQ). | Baseline and 14-weeks
Change in Medication Adherence as measured by Morisky Medication Adherence Scale (MMAS-8). | Baseline and 14-weeks
Change in Body Mass | Baseline and 14-weeks
  Weight
Change in Body Mass Index | Baseline and 14-weeks
  Weight/Height (kg/m2)
Change in waist circumference | Baseline and 14-weeks
  Minimal and Abdominal

CONTACTS AND LOCATIONS:
Overall Officials: William E Kraus, MD, Principal Investigator — Duke University
Locations (1):
- Duke Medicine - Duke Molecular Physiology Institute, Durham, North Carolina, United States

REFERENCES:
- [Derived] Duscha BD, Piner LW, Patel MP, Craig KP, Brady M, McGarrah RW 3rd, Chen C, Kraus WE. Effects of a 12-week mHealth program on peak VO2 and physical activity patterns after completing cardiac rehabilitation: A randomized controlled trial. Am Heart J. 2018 May;199:105-114. doi: 10.1016/j.ahj.2018.02.001. Epub 2018 Feb 7. PMID 29754647